CLINICAL TRIAL: NCT05391217
Title: Study to Remotely Monitor Activity in Transgender Cancer Survivors
Brief Title: Feasibility of Remote Activity Assessment and PRO Collection Among Transgender Cancer Survivors
Acronym: STRIDE
Status: Recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Gillian Gresham, Assistant Professor, Cedars-Sinai Medical Center
Other Study IDs: STUDY00001826
Record Dates: First submitted 2022-04-20; First posted 2022-05-25 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Neoplasms; Chronic Disease
MeSH Terms: conditions — Neoplasms; Chronic Disease | interventions — Activities of Daily Living

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transgender people with history of cancer: Self-reported cancer history and/or treatment for cancer within the last 5 years.
  Interventions: Other: Remote assessment of patient reported outcomes and daily activity
- Transgender people without history of cancer: People living with other chronic conditions
  Interventions: Other: Remote assessment of patient reported outcomes and daily activity

INTERVENTIONS:
Other: Remote assessment of patient reported outcomes and daily activity — Electronic patient-reported outcomes (NIH PROMIS) will be collected and combined with remotely monitored physical activity, heart rate, and sleep, as measured with a Fitbit (Sense).
  Other Names: PROs + remote physical activity monitoring

SUMMARY:
Prospective observational feasibility study to evaluate the role of wearable activity monitors to determine the feasibility and acceptability of remote monitoring using wearable technology and PROs to monitor fatigue and physical function in transgender cancer patients and survivors.

DETAILED DESCRIPTION:
Transgender cancer survivors are a diverse population who currently suffer from cancer-related disparities. Enrolled subjects will receive wearable activity devices to help understand how their daily activity (e.g., daily step counts, stairs climbed) and sleep levels are affected by their symptoms and treatment side-effects, including fatigue, physical functioning, emotional well-being, sleep quality, and quality of life over the 2-week course of the study. Qualitative interviews will be conducted to gain a deeper understanding of barriers to physical activity and their perceived relationships with their cancer history, treatment symptoms and gender affirming hormone therapy.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as transgender person with a history of cancer or receiving treatment for cancer in the last five years from screening for the current study (case) OR self-identifies as transgender person without a history of cancer (control)
* 18 years or older
* Ambulatory (use of walking aids, such as cane and rollator, is acceptable)
* Access to a device (e.g., smartphone, tablet, iPhone) that has the capability to sync to the Fitbit
* Have an understanding, ability, and willingness to fully comply with study procedures and restrictions
* Can read and understand English, Spanish, or Tagalog (for participant surveys and interviews)
* Informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Any person that does not meet the listed criteria above
* Using a pacemaker, implantable cardiac defibrillator, neurostimulator, implantable hearing aids, cochlear implants, or other electronic medical equipment*. However, removable hearing aids are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender man or woman, or identifies as transgender
Study Population: Self-identifies as transgender person with a history of cancer or receiving treatment for cancer in the last five years from screening for the current study (case) OR self-identifies as transgender person without a history of cancer (control)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Remote Activity Assessment and PRO Collection | 2 weeks
  Proportion of patients who consent to participate in the research study and complete the baseline fatigue assessment, where a proportion of 50% will be considered feasible.

SECONDARY OUTCOMES:
Key themes and concepts surrounding the relationships patients have with their treatment symptoms and how they affect their daily activity | 2 weeks
  Qualitative outcome, as obtained through semi-structured interviews
Average daily step count (steps/day) | 2 weeks
  Average daily step count over the study period will be calculated from wearable activity monitor
24-Hour Movement | 2 weeks
  A composite of average time spent in physical activity (light/moderate/vigorous), time sedentary, and sleep will be calculated following the 24-hour movement continuum guidelines and average values will be obtained over the study period.
Patient-reported health and well-being | 2 weeks
  NIH PROMIS surveys (Likert scale range 0-5, where 5 is the highest level of well-being) at baseline and end of study
Patient-reported mood | up to 2 weeks
  Mean NIH PROMIS anxiety, depression and stress scores (range 0-5), converted to T-scores (mean 50, SD 10) at each timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Gresham, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
This is a small feasibility trial with only 20 people from an underrepresented, minority population, thus important to maintain privacy and confidentiality.